CLINICAL TRIAL: NCT06413069
Title: Effects of Almonds in Glucose-intolerant Adults - a Randomised Controlled Study on Muscle Mass and Obesity, Energy Metabolism and Lipidome, NON-alcoholic Fatty Liver and Inflammation (AGAMEMNON)
Brief Title: Effects of Almonds in Glucose-intolerant Adults (AGAMEMNON)
Acronym: AGAMEMNON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Stefan Kabisch, Principal investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGAMEMNON
Record Dates: First submitted 2024-01-29; First posted 2024-05-14 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: PreDiabetes; NAFLD
Keywords: almonds; dietary treatment; diabetes prevention; metabolic syndrome
MeSH Terms: conditions — Prediabetic State; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: parallel, single-blinded, prospective, randomised controlled trial in waiting list design
Who Masked: Investigator, Outcomes Assessor
Masking Description: masking not possible; subjects are aware of their allocation after initiation of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond treatment (Active Comparator): Subjects will be supplemented with 60 grams of almonds (treatment) or left untreated (no-nut group) for 16 weeks.
  Interventions: Dietary Supplement: Raw whole almonds
- Control condition (No Intervention): Patients of the no-nut group will receive 6,7 kgs of almonds after completing 16 weeks of waiting time, supporting their compliance as untreated group.

INTERVENTIONS:
Dietary Supplement: Raw whole almonds — Subjects will be supplemented with 60 grams of almonds (treatment) or left untreated (no-nut group) for 16 weeks. Patients of the no-nut group will receive 6,7 kgs of almonds after finishing the study, supporting their compliance as untreated group.
  Arms: Almond treatment

SUMMARY:
Tree nuts - such as almonds - contribute to beneficial effects of the Mediterranean diet on risk for cardiovascular events, type 2 diabetes, dyslipidemia, hypertension, inflammation and non-alcoholic fatty liver disease. Almonds provide few carbohydrates, but lots of unsaturated fat and dietary fiber. But to which extent and by which mechanisms may almonds improve all aspects of the Metabolic Syndrome? Previous clinical trials showed weaker effects than rodent studies, most possibly due to low statistical power and metabolically insusceptible patients.

The 3-year AGAMEMNON project aims to investigate, if 16 weeks of supplementation with almonds (vs. no treatment) in 150 patients with prediabetes and NAFLD leads to significant improvements in glycemia and liver fat, lipid metabolism, body composition and inflammation. The isocaloric design will outrule effects of weight loss and will allow the analysis of metabolic pathways between fat depots, inflammation, insulin resistance and gut function. Lipidomics are assessed as novel predictor of disease progression and metabolic response.

DETAILED DESCRIPTION:
Background / Significance:

T2D affects 5-10 % of the global population, challenging societies, health systems, economy and quality of life. Dietary treatment may avoid disease burdens, save money and protect general health resources, but is often limited to unspecific weight loss recommendations and advise for physical activity. Despite being the common advice, body weight reduction is faced with inconclusive evidence for its impact on long-term risks (obesity paradox?), lack of long-term compliance and irresponsive or ineligible subgroups of patients. The Mediterranean diet provides the ideal dietary composition and reduces CVD risk, improving every axis of the Metabolic Syndrome, including liver fat. It is unclear, though, to which extent tree nuts contribute to this effect.

In meta-analyses, almonds improve glycemia and lipids. Benefits on body composition and inflammation are also expected, these might extend to NAFLD.

n6-PUFAs (typical components of tree nuts) reduce T2D risk and liver fat in humans. This was shown for sunflower oil, but not yet for nuts. Evidence for NAFLD benefits by almonds in humans is limited to observational studies, post-hoc analyses of mixed interventions, and underpowered RCTs.

Aims / Rationale:

Nuts are safe for NAFLD patients. Previous data indicate, that almonds may elicit benefits on glycemia and liver fat in patients susceptible to this treatment.

Therefore, the investigators' project aims to investigate whole almonds as dietary treatment for glucose intolerance and NAFLD in patients with this typical combined phenotype. NAFLD independently predicts T2D progression and late complications. (Pre)diabetes patients with NAFLD are at higher risk for the entire metabolic syndrome and for early onset of nephropathy and CVD. On the other hand, prediabetes/T2D patients with NAFLD are also especially susceptible to lifestyle treatments. The investigators hypothesize to detect benefits of almonds with respect to glycemia and liver fat, but also lipid metabolism, body composition and inflammation compared to standard diet. Treatment period of 16 weeks is longer than earlier almond studies.

The investigators intend to show, that the metabolic improvement is independent from weight loss and, even in the opposite, supports maintenance of muscle mass. The research group wants to investigate mechanistic links between the metabolic pathways of visceral fat accumulation, inflammation, NAFLD, insulin resistance, dyslipidemia and the gut microbiome. Finally, the investigators aim to assess the lipidome (analysed from the erythrocyte membranes, full blood and plasma samples), which was recently established as a novel biomarker to predict disease progression, metabolic response and treatment-specific improvement.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes (IFG or IGT or IFG-IGT), measured in plasma samples
* NAFLD (MR-S: >5,56 %)
* BMI between 25 and 40 kg/m²

Exclusion Criteria:

* Treatment with antidiabetic drugs
* Overt diabetes mellitus of any kind
* Severe cardiovascular or pulmonary disorder
* Renal disorder / Renal insufficiency (eGFR < 60 ml/min/m²)
* Severe psychiatric disorder (schizophrenia, severe depression; eating disorders)
* Current or recent (< 5 years) cancer diagnosis
* Liver disease other than NAFLD
* Use of corticosteroid treatments
* Alcohol abuse
* Smoking
* Ongoing or recently finished (3 months before) weight loss
* Current participation in other intervention studies
* Pregnancy
* Metal implants, claustrophobia
* Allergy to almonds

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Liver fat content | 16 weeks
  change in liver fat content (magnetic resonance spectroscopy)
concentration of fasting plasma glucose | 16 weeks
  change in concentration of fasting plasma glucose
concentration of 2-h plasma glucose (75 g oGTT) | 16 weeks
  change in concentration of 2-h plasma glucose (75 g oGTT)

SECONDARY OUTCOMES:
whole body fat content (%; measured with BIA) | 16 weeks
  change in whole body fat content
whole body fat content (kg; measured with BIA) | 16 weeks
  change in whole body fat content
insulin sensitivity (Matsuda) | 16 weeks
  change in insulin sensitivity (Matsuda)
insulin secretion capacity (disposition index-2); metric parameter without defined maxima or minima; higher values indicate better insulin secretion | 16 weeks
  change in insulin secretion capacity (disposition index-2); metric parameter without defined maxima or minima; higher values indicate better insulin secretion
blood pressure (sys/dia) | 16 weeks
  change in blood pressure (sys/dia)
serum concentration of CRP | 16 weeks
  change in serum concentration of CRP
serum concentration of IL-6 | 16 weeks
  change in serum concentration of IL-6
serum concentration of IL-10 | 16 weeks
  change in serum concentration of IL-10
serum concentration of IL-1ß | 16 weeks
  change in serum concentration of IL-1ß
serum concentration of IL-18 | 16 weeks
  change in serum concentration of IL-18
serum concentration of IL-22 | 16 weeks
  change in serum concentration of IL-22
fasting triglyceride levels | 16 weeks
  change in fasting triglyceride levels
LDL, HDL, LDL/HDL ratio | 16 weeks
  change in LDL, HDL, LDL/HDL ratio
concentration of serum lipidome parameters (hundreds of lipid species) | 16 weeks
  change in serum lipidome (hundreds of lipid species)

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University Hospital Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided